CLINICAL TRIAL: NCT02828345
Title: Bio-marker Analysis Using Circulating Tumor Cells in Patients With Melanoma
Status: Withdrawn | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15613
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Specimen Collection

SUMMARY:
This research trial studies the levels of a type of biomarker, circulating tumor cells (CTCs), in the blood of patients with stage I-IV melanoma. A biomarker is a biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition. Studying samples of blood in the laboratory obtained before and after treatment from patients with melanoma may help doctors learn more about changes that occur in CTC levels and whether they may predict how well patients will respond to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed tissue collection consent as described in protocol IRB# 703001,UPCC# 08607, PI: Giorgos Karakousis, MD
* Subjects must be competent to consent for themselves.
* Subjectsmust be adult (18 years or older).
* Subjects must be initiating a new therapy for melanoma (so a pretreatment CTC count can be obtained).

Exclusion Criteria:

* Children (less than 18yrs)
* Patients in whom a pre-treatment CTC level cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Melanoma
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of changes in CTC level from pre- to post-treatment | two years

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Karakousis, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine